CLINICAL TRIAL: NCT06473779
Title: A Multicentre, Randomised, Open-Label, Parallel-Group, Phase IIIb Study to Assess the Potential for Tezepelumab-treated Patients With Severe Asthma to Reduce Background Therapy While Sustaining Asthma Control and Clinical Remission
Brief Title: Open-label Study to Assess Reduction of Background Asthma Medication While Sustaining Asthma Control and Clinical Remission With Tezepelumab in Patients 12-80yrs With Severe Asthma.
Acronym: ARRIVAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5180C00047
Record Dates: First submitted 2024-06-10; First posted 2024-06-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Severe Asthma
Keywords: Severe Asthma; ICS reduction; Asthma control; Clinical remission
MeSH Terms: conditions — Asthma | interventions — tezepelumab; Budesonide, Formoterol Fumarate Drug Combination; Albuterol; Budesonide; Mannitol

STUDY DESIGN:
Intervention Model Description: Open-Label, Parallel-Group treatment study with 3 arms. Participants will be treated with tezepelumab Q4W from Week 0, with the last dose administered at Week 68
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Group 1 - Asthma Control or Low Biomarkers - Step-down of ICS (Experimental): Asthma Control or Low Biomarkers - Step-down of ICS. Only patients with asthma control or low biomarkers at Week 24 will be randomized into Group 1 or 2
  Interventions: Combination Product: Tezepelumab; Combination Product: Budesonide/formoterol; Combination Product: Albuterol/budesonide (AIRSUPRA®); Combination Product: Mannitol; Combination Product: Salbutamol
- Group 2 - Asthma Control or Low Biomarkers - No Step-down of ICS (Experimental): Asthma Control or Low Biomarkers - No Step-down of ICS. Only patients with asthma control or low biomarkers at Week 24 will be randomized into Group 1 or 2
  Interventions: Combination Product: Tezepelumab; Combination Product: Budesonide/formoterol; Combination Product: Albuterol/budesonide (AIRSUPRA®); Combination Product: Mannitol; Combination Product: Salbutamol
- Group 3 - No Asthma Control or Low Biomarkers - No Step-down of ICS (Experimental): No Asthma Control or Low Biomarkers - No Step-down of ICS
  Interventions: Combination Product: Tezepelumab; Combination Product: Budesonide/formoterol; Combination Product: Albuterol/budesonide (AIRSUPRA®); Combination Product: Mannitol

INTERVENTIONS:
Combination Product: Tezepelumab — IMP. Subcutaneous injection. Unit dose strengths 210 mg.
  Other Names: TEZSPIRE®
Combination Product: Budesonide/formoterol — AxMP. Oral inhalation. High-dose: 160 μg/4.5 μg per inhalation; Medium and Low-dose: 80 μg/4.5 μg per inhalation
  Other Names: SYMBICORT® pMDI
Combination Product: Albuterol/budesonide (AIRSUPRA®) — AxMP. Oral inhalation. Reliever only. Unit dose strengths 90 μg/80 μg per inhalation In US only.
  Other Names: AIRSUPRA®
Combination Product: Mannitol — NIMP. Oral nebulization. Unit dose strengths: Graduated doses of 0 mg, 5 mg, 10 mg, 20 mg and 40 mg capsules
  Other Names: ARIDOL®
Combination Product: Salbutamol — AxMP. Used outside the US only. Oral inhalation. Unit dose strengths: 100 μg per inhalation
  Other Names: Sabumalin, albuterol, ventolin HFA, Proair HFA, Proventil HFA
  Arms: Group 1 - Asthma Control or Low Biomarkers - Step-down of ICS; Group 2 - Asthma Control or Low Biomarkers - No Step-down of ICS

SUMMARY:
The objective of this study is to assess the potential for tezepelumab-treated patients (subcutaneous administration) to reduce maintenance therapy without loss of asthma control in adolescent and adults with severe asthma..

Study details include:

1. The study duration will be up to 72 weeks.
2. The treatment duration will be up to 68 weeks.
3. The visit frequency will be once every 4 weeks (Q4W).

DETAILED DESCRIPTION:
This is a multicentre, randomised, open-label, parallel-group, phase IIIb study to assess the potential for tezepelumab-treated patients to (1) reduce maintenance therapy without the loss of asthma control at Week 56, among those who demonstrated asthma control or low biomarkers at Week 24, and (2) be in asthma control and have characteristics of clinical remission at Week 24.

Approximately 65 sites in 10 countries will enrol adult and adolescent patients with severe uncontrolled asthma.

The study is divided into 5 phases as described below:

* Screening/Run-in Phase (from Week -4 until Week 0, up to 4 Weeks)
* Treatment Induction Phase (Week 0 to Week 4)
* Treatment Continuation Phase (Week 4 to Week 24)
* Tezepelumab Treatment With or Without ICS Step-down Therapy Phase (Week 24 to Week 56)
* Maintenance Phase (Week 56 to Week 72)

ELIGIBILITY:
Inclusion Criteria at Visit 1 (Screening):

Informed Consent

1. Provision of signed and dated written ICF prior to any mandatory study-specific procedures, sampling, and analyses for patients who are at or over the age of majority (as per local law). For patients who are less than the age of majority, in addition to providing their informed consent, the patients' legally authorised representative must also provide their informed assent (Appendix A 3).

   Age
2. Patients must be 12 to 80 years of age inclusive, at the time of signing the ICF.

   Type of Patient and Disease Characteristics
3. Documented medical record history for at least 12 months prior to Visit 1.
4. Documented physician-diagnosed severe asthma within 10 years prior to Visit 1 (ie, severe asthma was not diagnosed more than 10 years prior) consisting of any of the following:

   1. FEV1 > 12% reversibility, OR
   2. Evidence of airflow variability (to show that lung function is altered over time): FEV1 ≥ 400 mL variability over time, OR
   3. Challenge tests that are positive on one of the below:

   (i) Methacholine - PD20 ≤ 8 mg/mL (ii) Mannitol - PD15 15% drop on FEV1 out of dose < than 635 mg of inhaled mannitol (iii) Exercise - 10% fall of FEV1
5. ACQ-5 ≥ 1.5 and < 3.
6. History of physician-diagnosed asthma that requires continuous treatment with high-dose ICS (as defined by GINA or highest approved dose per posology per country) plus a LABA for at least 6 months prior to Visit 1 (Appendix I). The ICS and LABA can be contained within a combination product or given by separate inhalers.

   Note: Additional maintenance asthma controller medications (eg, LTRAs, tiotropium, cromone, theophylline) are allowed.
7. Pre-brochodilator FEV1 > 60% predicted and evidence of FEV1 reversibility of > 12% within 6 months prior to screening or at screening. Patients with normal lung function (FEV1 > 80%) need evidence of airflow variability as per inclusion criterion 4.
8. Documented history of at least one asthma exacerbation requiring OCS bursts or requiring hospitalization within 12 months prior to Visit 1. An asthma exacerbation will be defined as a worsening of asthma symptoms that leads to any of the following:

   1. A temporary bolus/burst of systemic corticosteroids for at least 3 consecutive days to treat symptoms of asthma worsening; a single depo-injectable dose of corticosteroids will be considered equivalent to a 3-day bolus/burst of systemic corticosteroids
   2. Or, an ER visit (defined as evaluation and treatment for < 24 hours in ER) due to asthma that required systemic corticosteroids (as per above)
   3. Or, an in-patient hospitalisation (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥ 24 hours).

   Sex and Contraceptive/Barrier Requirements
9. Male or female.

   Female patients:
   * Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Women of nonchildbearing potential are defined as women who are either permanently sterilised (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to the planned start date of the induction phase without an alternative medical cause.
   * The following age-specific requirements apply:

     * Women < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and follicle-stimulating hormone levels in the postmenopausal range.
     * Women ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatment.
     * Adolescents: if patient is female and has reached menarche or has reached Tanner stage 3 breast development (even if not having reached menarche), the patient will be considered a WOCBP.
10. WOCBP must be willing to use one of the methods of contraception described hereafter, from the time of signing the ICF throughout the study and 16 weeks after last tezepelumab administration:

    * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: oral, intravaginal, transdermal
    * Progestogen-only hormonal contraception associated with inhibition of ovulation: oral, injectable, implantable
    * Intrauterine device
    * Intrauterine hormone-releasing system
    * Bilateral tubal occlusion
    * Vasectomised partner (vasectomised partner is a highly effective birth control method provided that the partner is the sole sexual partner of the WOCBP patient and that the vasectomised partner has received medical assessment of the surgical success)
    * Sexual abstinence: it is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient.
    * Cessation of contraception after this point should be discussed with a responsible physician

    Inclusion Criteria 5.1.2 Treatment Induction Phase at Visit 2 (Week 0):

    Before dosing with tezepelumab at Week 0, patients should fulfil the following criteria:
11. ACQ-5 ≥ 1.5 and < 3.
12. Demonstrated proper inhaler technique (patients with improper technique at screening may be trained during screening, but must demonstrate proper technique before enrollment).
13. No excessive SABA use (should be < 5 puffs/day) or for patients using SMART therapy outside the US, no excessive use of SYMBICORT (should be ≤ 8 inhalations/day) or for US patients, no excessive use of AIRSUPRA (should be ≤ 12 inhalations/day).

Exclusion Criteria:

Medical Conditions

1. Any clinically important pulmonary disease other than asthma (eg, active lung infection, chronic obstructive pulmonary disease, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or pulmonary or systemic diseases, other than asthma, that are associated with elevated peripheral EOS counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
2. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the study or the interpretation
   * Impede the patient's ability to complete the entire duration of study.
3. A helminth parasitic infection diagnosed within 6 months prior to Visit 1 that has not been treated with, or has failed to respond to, standard of care therapy.
4. Current smokers or patients with smoking history ≥ 10 pack-years and patients using vaping products, including electronic cigarettes. Former smokers with a smoking history of < 10 pack-years and users of vaping or e-cigarette products must have stopped for at least 6 months prior to Visit 1 to be eligible.
5. History of chronic alcohol or drug abuse within 12 months prior to Visit 1.
6. Tuberculosis requiring treatment within the 12 months prior to Visit 1.
7. History of known immunodeficiency disorder including a positive human immunodeficiency virus test at Visit 1, or the patient taking antiretroviral medications as determined by medical history and/or patient's verbal report.
8. Major surgery within 8 weeks prior to Visit 1 or planned surgical procedures requiring general anaesthesia or inpatient status for > 1 day during the conduct of the study.
9. Evidence of COVID-19 within 4 weeks prior to screening or ongoing clinically significant COVID-19 sequelae.

   Prior/Concomitant Therapy
10. Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives (whichever is longer) prior to Visit 1 or receipt of any investigational nonbiologic agent within 30 days or 5 half-lives (whichever is longest) prior to Visit 1.
11. OCS-dependent patients (received chronic OCS therapy [prednisone ≥ 5 mg/day or equivalent]) for at least 3 months preceding Visit 1.
12. Daily use of maintenance corticosteroids for any reason.
13. Treatment with systemic immunosuppressive/immunomodulating drugs (eg, methotrexate, cyclosporine, etc.), except for OCS used in the treatment of asthma/asthma exacerbations, within the last 12 weeks or 5 half-lives (whichever is longer) prior to Visit 1.
14. Receipt of immunoglobulin or blood products within 30 days prior to Visit 1.
15. Receipt of live attenuated vaccines 30 days prior to the date of Visit 1 and during the study.
16. Patients that have been treated with bronchial thermoplasty in the last 12 months prior to Visit 1.

    Prior/Concurrent Clinical Study Experience
17. Known history of sensitivity to any component of the tezepelumab formulation or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
18. History of anaphylaxis or documented immune complex disease (Type III hypersensitivity reactions) following any biologic therapy.
19. Concurrent enrolment in another clinical study involving an IMP.

    Diagnostic Assessments
20. Any clinically meaningful abnormal finding in physical examination, haematology, clinical chemistry at Visit 1 which, in the opinion of the investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete the entire duration of the study.
21. Evidence of active liver disease, including jaundice or AST, ALT, or ALP > 2 times the ULN at Visit 1.
22. Positive hepatitis B surface antigen, hepatitis C virus antibody serology at screening, or a positive medical history for hepatitis B or C. Patients with a history of hepatitis B vaccination without a history of hepatitis B are allowed to participate.

    Other Exclusions
23. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or site staff), or patients employed by or relatives of the employees of the site or AstraZeneca.
24. Judgement by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
25. For women only: Pregnant, breastfeeding, or lactating women. A serum β-HCG pregnancy test must be drawn for WOCBP at the screening visit. If the results of the serum β-HCG cannot be obtained prior to dosing of the IMP, a patient may be enrolled on the basis of a negative urine pregnancy test, though serum β-HCG must still be obtained. If either test is positive, the patient should be excluded. Since urine and serum tests may miss a pregnancy in the first days after conception, relevant menstrual history and sexual history, including methods of contraception, should be considered. Any patient whose menstrual and/or sexual history suggests the possibility of early pregnancy should be excluded.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who reduced their SYMBICORT® daily maintenance dose without the loss of asthma control at the end of the step-down phase. | Week 56
  Proportion of patients who reduced their SYMBICORT® daily maintenance dose without the loss of asthma control at the end of the step-down phase to either:
  Outside of the US:
  * Medium-dose maintenance and reliever therapy, or
  * Low-dose maintenance and reliever therapy, or
  * SYMBICORT® anti-inflammatory reliever only
  In the US:
  * Medium-dose SYMBICORT® and AIRSUPRA®,or
  * Low-dose SYMBICORT® and AIRSUPRA®, or
  * AIRSUPRA® only

SECONDARY OUTCOMES:
Proportion of patients in asthma control | Week 24
  Proportion of patients in asthma control at Week24.
Proportion of patients with characteristics of clinical remission | Week 24
  Proportion of patients with characteristics of clinical remission at Week 24
Proportion of patients in asthma control at Week 56 among those in asthma control at Week 24 | Week 56
  Proportion of patients in asthma control at Week 56 among those in asthma control at Week 24; summarised separately for patients randomised to ICS step-down and for patients randomised to no step-down of ICS.
Proportion of patients in asthma control at Week 72 among those in asthma control at Week 24 | Week 72
  Proportion of patients in asthma control at Week 72 among those in asthma control at Week 24; summarised separately for patients randomised to ICS step-down and for patients randomised to no step-down of ICS.
Proportion of patients in asthma control at both Week 56 and Week 72 among those in asthma control at Week 24 | Week 56 and Week 72
  Proportion of patients in asthma control at both Week 56 and Week 72 among those in asthma control at Week 24; summarised separately for patients randomised to ICS step-down and for patients randomised to no step-down of ICS.
Proportion of patients in asthma control at Week 56 among those who demonstrated neither asthma control nor low biomarkers at Week 24 | Week 56
  Proportion of patients in asthma control at Week 56 among those who demonstrated neither asthma control nor low biomarkers at Week 24
Proportion of patients in asthma control at Week 72 among those who demonstrated neither asthma control nor low biomarkers at Week 24 | Week 72
  Proportion of patients in asthma control at Week 72 among those who demonstrated neither asthma control nor low biomarkers at Week 24
Proportion of patients in clinical remission at Week 56 among those with characteristics of clinical remission at Week 24 | Week 56
  Proportion of patients in clinical remission at Week 56 among those with characteristics of clinical remission at Week 24; summarised separately for patients randomised to ICS step-down and for patients randomised to no step-down of ICS.
Proportion of patients in clinical remission at Week 72 among those with characteristics of clinical remission at Week 24 | Week 72
  Proportion of patients in clinical remission at Week 72 among those with characteristics of clinical remission at Week 24; summarised separately for patients randomised to ICS step-down and for patients randomised to no step-down of ICS.
Proportion of patients in clinical remission at both Week 56 and Week 72 among those with characteristics of clinical remission at Week 24 | Week 56 and Week 72
  Proportion of patients in clinical remission at both Week 56 and Week 72 among those with characteristics of clinical remission at Week 24; summarised separately for patients randomised to ICS step-down and for patients randomised to no step-down of ICS.
Proportion of patients in clinical remission at Week 56 among those who demonstrated neither asthma control nor low biomarkers at Week 24 | Week 56
  Proportion of patients in clinical remission at Week 56 among those who demonstrated neither asthma control nor low biomarkers at Week 24
Proportion of patients in clinical remission at Week 72 among those who demonstrated neither asthma control nor low biomarkers at Week 24 | Week 72
  Proportion of patients in clinical remission at Week 72 among those who demonstrated neither asthma control nor low biomarkers at Week 24
Proportion of patients in complete remission at Week 56 | Week 56
  Proportion of patients in complete remission at Week 56; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Proportion of patients in complete remission at Week 72 among those in complete remission at Week 56 | Week 72
  Proportion of patients in complete remission at Week 72 among those in complete remission at Week 56; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Change from Week 24 at Week 56 in: ° Mean monthly maintenance ICS dose ° Mean monthly rescue ICS dose ° Mean monthly total ICS dose (maintenance and rescue doses) | From Week 24 at Week 56
  Change from Week 24 at Week 56 in:
  * Mean monthly maintenance ICS dose
  * Mean monthly rescue ICS dose
  * Mean monthly total ICS dose (maintenance and rescue doses)
Change from Week 24 at Week 72 in: ° Mean monthly maintenance ICS dose ° Mean monthly rescue ICS dose ° Mean monthly total ICS dose (maintenance and rescue doses) | From Week 24 at Week 72
  Change from Week 24 at Week 72 in:
  * Mean monthly maintenance ICS dose
  * Mean monthly rescue ICS dose
  * Mean monthly total ICS dose (maintenance and rescue doses)
Cumulative daily ICS dose (maintenance and rescue doses) between Week 24 and Week 56 | Between Week 24 and Week 56
  Cumulative daily ICS dose (maintenance and rescue doses) between Week 24 and Week 56 both summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Cumulative daily ICS dose (maintenance and rescue doses) between Week 56 and Week 72 | Between Week 56 and Week 72
  Cumulative daily ICS dose (maintenance and rescue doses) between Week 56 and Week 72 both summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Cumulative daily ICS dose (maintenance and rescue doses) between Week 24 and Week 72 | Between Week 24 and Week 72
  Cumulative daily ICS dose (maintenance and rescue doses) between Week 24 and Week 72 both summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
AAER between Week 0 and Week 24 among all tezepelumab-treated patients | Between Week 0 and Week 24
  Annualised Asthma Exacerbation Rate between Week 0 and Week 24 among all tezepelumab-treated patients.
AAER between Week 24 and Week 56 | Between Week 24 and Week 56
  Annualised Asthma Exacerbation Rate between Week 24 and Week 56 summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
AAER between Week 56 and Week 72 | Between Week 56 and Week 72
  Annualised Asthma Exacerbation Rate between Week 56 and Week 72 summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
AAER between Week 24 and Week 72 | Between Week 24 and Week 72
  Annualised Asthma Exacerbation Rate between Week 24 and Week 72 summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
ACQ-5 score and changes from baseline at Week 24 among all tezepelumab-treated patients | From baseline at Week 24
  ACQ-5 score and changes from baseline at Week 24 among all tezepelumab-treated patients
ACQ-5 score and changes from Week 24 at Week 56 | From Week 24 at Week 56
  ACQ-5 score and changes from Week 24 at Week 56; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
ACQ-5 score and changes from Week 24 at Week 72 | From Week 24 at Week 72
  ACQ-5 score and changes from Week 24 at Week 72; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Proportion of ACQ-5 responders (improvement of≥ 0.5 in ACQ-5 score) from baseline at Week 24 among all tezepelumab-treated patients. | From baseline at Week 24
  Proportion of ACQ-5 responders (improvement of≥ 0.5 in ACQ-5 score) from baseline at Week 24 among all tezepelumab-treated patients.
Proportion of ACQ-5 responders (improvement of≥ 0.5 in ACQ-5 score) from Week 24 at Week 56 | From Week 24 at Week 56
  Proportion of ACQ-5 responders (improvement of≥ 0.5 in ACQ-5 score) from Week 24 at Week 56; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Proportion of ACQ-5 responders (improvement of≥ 0.5 in ACQ-5 score) from Week 24 at Week 72 | From Week 24 at Week 72
  Proportion of ACQ-5 responders (improvement of≥ 0.5 in ACQ-5 score) from Week 24 at Week 72; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
SGRQ total score and changes from baseline at Week 24 among all tezepelumab-treated patients. | From baseline at Week 24
  SGRQ total score and changes from baseline at Week 24 among all tezepelumab-treated patients.
SGRQ total score and changes from Week 24 at Week 56 | From Week 24 at Week 56
  SGRQ total score and changes from Week 24 at Week 56, summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
SGRQ total score and changes from Week 24 at Week 72 | From Week 24 at Week 72
  SGRQ total score and changes from Week 24 at Week 72, summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Proportion of SGRQ responders (improvement of≥ 4 in SGRQ total score) from baseline at Week 24 among all tezepelumab-treated patients. | From baseline at Week 24
  Proportion of SGRQ responders (improvement of≥ 4 in SGRQ total score) from baseline at Week 24 among all tezepelumab-treated patients
Proportion of SGRQ responders (improvement of≥ 4 in SGRQ total score) from Week 24 at Week 56 | From Week 24 at Week 56
  Proportion of SGRQ responders (improvement of≥ 4 in SGRQ total score) from Week 24 at Week 56; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Proportion of SGRQ responders (improvement of≥ 4 in SGRQ total score) from Week 24 at Week 72 | From Week 24 at Week 72
  Proportion of SGRQ responders (improvement of≥ 4 in SGRQ total score) from Week 24 at Week 72; summarised separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Pre-BD FEV1 actual values and changes from baseline at Week 24 among all tezepelumab-treated patients. | Baseline at Week 24
  Asthma exacerbations, patient-reported outcomes, and lung function. Pre-BD FEV1 actual values and changes from baseline at Week 24 among all tezepelumab-treated patients.
Pre-BD FEV1 total score and changes from Week 24 at Week 56 | From Week 24 at Week 56
  Pre-BD FEV1 total score and changes from Week 24 at Week 56, summarized separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24 among all tezepelumab-treated patients.
Pre-BD FEV1 total score and changes from Week 24 at Week 72 | From Week 24 at Week 72
  Pre-BD FEV1 total score and changes from Week 24 at Week 72, summarized separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24 among all tezepelumab-treated patients.
Proportion of pre-BD FEV1 responders from baseline at Week 24 | Week 24
  Proportion of pre-BD FEV1 responders from baseline (defined as patients who achieve either a≥ 5% or ≥ 100 mL improvement from baseline) at Week 24, for all tezepelumab-treated patients
Proportion of pre-BD FEV1 responders at Week 56 among those who were pre-BDFEV1 responders at Week 24 | Week 56
  Proportion of pre-BD FEV1 responders at Week 56 among those who were pre-BDFEV1 responders at Week 24; summarized separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.
Proportion of pre-BD FEV1 responders at Week 72 among those who were pre-BDFEV1 responders at Week 24 | Week 72
  . Proportion of pre-BD FEV1 responders at Week 72 among those who were pre-BDFEV1 responders at Week 24; summarized separately for patients randomised to ICS step-down, randomised to no ICS step-down, and those who demonstrated neither asthma control nor low biomarkers at Week 24.

CONTACTS AND LOCATIONS:
Locations (64):
- United States (8):
  - Research Site, Palmdale, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Miami, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, New Brunswick, New Jersey
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, McAllen, Texas
- Argentina (8):
  - Research Site, Berazategui
  - Research Site, CABA
  - Research Site, Concepción del Uruguay
  - Research Site, Mendoza
  - Research Site, Quilmes
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Belgium (5):
  - Research Site, Anderlecht
  - Research Site, Edegem
  - Research Site, Erpent
  - Research Site, Ghent
  - Research Site, Liège
- Bulgaria (7):
  - Research Site, Haskovo
  - Research Site, Pleven
  - Research Site, Razgrad
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Velika Tarnovo
- Canada (6):
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Regina, Saskatchewan
- Denmark (4):
  - Research Site, Aalborg
  - Research Site, Hvidovre
  - Research Site, Svendborg
  - Research Site, Vejle
- France (6):
  - Research Site, Créteil
  - Research Site, La Tronche
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Strasbourg
- Germany (5):
  - Research Site, Augsburg
  - Research Site, Bonn
  - Research Site, Cottbus
  - Research Site, Hanover
  - Research Site, Mainz
- Italy (4):
  - Research Site, Florence
  - Research Site, Orbassano
  - Research Site, Roma
  - Research Site, Verona
- Mexico (3):
  - Research Site, Chihuahua City
  - Research Site, Cuauhtémoc
  - Research Site, Monterrey
- Spain (4):
  - Research Site, Badalona(Barcelona)
  - Research Site, Barcelona
  - Research Site, Lugo
  - Research Site, Madrid
- United Kingdom (4):
  - Research Site, Belfast
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/